CLINICAL TRIAL: NCT04040881
Title: Accuracy of a Mobile Sensor-Based System for the Detection of Chemotherapy Toxicity in Older Adults With Cancer in a Developing Country
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GER-3037-19-22-1
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Older adults; Smartphones; eHealth; mHealth; Remote monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote monitoring using Smartphone (Experimental): Patients will be provided with a Global System for Mobile communications (GSM) accelerometer-equipped Android smartphone (specific model to be decided) with an installed open source, freely available pedometer application (Google Fit, Google, CA, United States) which will record their daily steps. Patients will receive daily calls from a research assistant to document the presence of clinically significant chemotherapy-related toxicity.
  Interventions: Behavioral: Remote monitoring using smartphone accelerometer

INTERVENTIONS:
Behavioral: Remote monitoring using smartphone accelerometer — Patients will be instructed to carry the smartphone around their hips during waking hours, regardless of whether they are at home or outside (a nylon hip holster will be provided) and to keep it turned on at all times.
  Daily steps will be recorded for at least seven days before the start of chemotherapy, and the median baseline number of daily steps will be calculated for each patient.
  On the first day of chemotherapy, patients will receive side effect education as per standard of care. Patients will be instructed to continue carrying the smartphone daily as indicated for the entire duration of the first three chemotherapy cycles.
  At the end of the follow-up period (or sooner in cases of early interruption of chemotherapy due to toxicity or disease progression; a change in chemotherapy regimen; or hospitalizations lasting ≥3 days), patients will rate their satisfaction with the intervention using a Likert-scale questionnaire and open-ended questions.

SUMMARY:
Patients with cancer in developing countries face considerable challenges in obtaining access to care due to a lack of human resources and infrastructure. This is particularly pressing for vulnerable populations such as older adults. In this setting, many patients receiving chemotherapy are unable to report the presence of toxicities, and adverse events can go unnoticed for considerable amounts of time. The goal of this study is to assess the accuracy of an objective patient-centered measure of physical function (the number of steps taken per day measured using an accelerometer-equipped smartphone) for the remote detection of chemotherapy toxicity in older adults. This study builds on a pilot trial showing that monitoring older patients remotely utilizing an accelerometer-equipped smartphone is feasible and acceptable, and that a decline in the number of steps detected using the device can be an early sign of chemotherapy toxicity. The hypothesis of this study is that a decline in the number daily steps from a prechemotherapy baseline, measured using an accelerometer-equipped smartphone, will be accurate for detecting chemotherapy toxicity in older adults with cancer. This study will evaluate the ability of a patient-centered measure (a decline in the number of daily steps compared with a pre-chemotherapy baseline) to identify the presence of clinically-significant chemotherapy-related toxicity in Mexican older adults with cancer starting first line chemotherapy. Patients will be provided with an accelerometer-equipped smartphone with an installed pedometer application. Baseline steps per day will be obtained and recorded before starting chemotherapy. The patients' steps will be monitored daily for the first three chemotherapy cycles and compared with baseline recordings. Patients will be contacted daily and chemotherapy toxicity will be assessed by a physician. If significant toxicities are identified, the patient will be prompted to seek medical attention. The optimal cutoff point for detecting chemotherapy toxicity utilizing a decline in the number of daily steps will be chosen and validated. The adherence and satisfaction with the intervention will also be evaluated. This study could improve current methods and transform the way in which cancer care is delivered by demonstrating that a simple patient-centered measure obtained using a commercially available smartphone can aid in the accurate identification of clinically significant toxicities among a vulnerable population such as older adults with cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* Any solid tumor
* Starting first-line chemotherapy
* Adjuvant, metastatic or recurrent setting
* Any socioeconomic and educational level

Exclusion Criteria:

* Patients with walking disability
* Bedridden patients (ECOG 3)
* Second or subsequent line of chemotherapy
* Inpatients
* Patients receiving radiation concomitantly with chemotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Accuracy | Three months
  We will determine the diagnostic accuracy of percent decline in daily steps (index test) for detecting patient (pt) reported chemotherapy (CT) toxicity (Tox) (reference standard) using the area under the curve (AUC) of the receiver operating characteristic (ROC) curve.

SECONDARY OUTCOMES:
Adherence | Three months
  Ratio of the number of days steps are uploaded (X) to the number of days (N) the pt was asked to carry the phone, reported as a percentage (X/N x100).
Patient Satisfaction | Three months
  Percentage of pts reporting a high satisfaction with their experience carrying the smartphone

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Soto Pérez de Celis, MD,MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No